CLINICAL TRIAL: NCT06936371
Title: Evaluation of the Effects of Open Bite Activator and Anterior Skeletal Anchorage-Supported Vertical Elastics on Dentofacial Structures in Skeletal Open Bite Cases
Brief Title: Treatment of Skeletal Open Bite With Open Bite Activator and Skeletal Anchorage-Supported Vertical Elastics
Acronym: SOBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Murat Kaan Erdem, Assistant Professor, Ankara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUFDT-ORT-2021-22; 36290600/22 (Other: Ankara University Faculty of Dentistry Clinical Research Ethics Committee)
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Skeletal Open Bite; Vertical Maxillary Excess; Hyperdivergent Growth Pattern; Long Face Syndrome
Keywords: Open Bite Activator; Skeletal Anchorage; Mini-screws; Vertical Elastics; Orthodontic Treatment; Anterior Open Bite; Bite Correction; Dentofacial Effects; Cephalometric Analysis; Growing Patients; Non-extraction Treatment; Functional Appliance; Vertical Dimension Control

STUDY DESIGN:
Intervention Model Description: This prospective interventional study employed a single-group design where all participants received the same treatment protocol: open bite activator combined with skeletal anchorage-supported vertical elastics. Participants were evaluated at baseline (T0) and after 12 months of treatment (T1).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional Appliance and Skeletal Anchorage Group (Experimental): This arm includes growing individuals with skeletal open bite treated using a combination of an open bite activator (functional appliance) and vertical intermaxillary elastics supported by anterior skeletal anchorage (mini-screws placed between lateral and canine teeth in both jaws). The appliance was worn full-time for 12 months. Cephalometric changes were evaluated before and after treatment to assess skeletal and dentoalveolar effects without the use of extraoral appliances.
  Interventions: Device: Open Bite Activator with Skeletal Anchorage-Supported Vertical Elastics

INTERVENTIONS:
Device: Open Bite Activator with Skeletal Anchorage-Supported Vertical Elastics — Participants received a removable open bite activator constructed with the mandible opened beyond the freeway space and combined with vertical intermaxillary elastics applying 150g of force, supported by mini-screws placed between the lateral and canine teeth in both the maxilla and mandible. The appliance was worn 20-22 hours daily for 12 months. This approach aimed to treat skeletal open bite without using extraoral appliances by promoting anterior mandibular rotation and inhibiting posterior vertical dentoalveolar development.
  Other Names: Functional Appliance with Mini-screw-Supported Elastics; Anterior Skeletal Anchorage

SUMMARY:
This study evaluated a new treatment approach for skeletal open bite in growing individuals using an open bite activator combined with anterior skeletal anchorage-supported vertical elastics. An open bite is a condition where the front teeth don't touch when the back teeth are closed together, creating a gap. Traditional treatments often use extraoral appliances (devices worn outside the mouth), which can be uncomfortable and aesthetically unappealing, leading to poor patient compliance.

We included 24 growing patients (14 females, 10 males) aged 12-14 years with skeletal open bite. All participants received an open bite activator (a removable functional appliance) and mini-screws placed between the upper and lower lateral and canine teeth. Vertical elastics were connected between these mini-screws, applying 150g of force for 20-22 hours daily over 12 months.

Lateral cephalometric radiographs (specialized X-rays) were taken before treatment and after 12 months to evaluate changes in facial bone structure and tooth positions. Our results showed successful correction of open bite with an average increase in overbite of 3.35mm. We observed favorable skeletal changes including clockwise rotation of the maxilla (upper jaw), counterclockwise rotation of the mandible (lower jaw), and decreased vertical facial dimensions.

This treatment approach offers a viable alternative to conventional methods that rely on extraoral appliances, potentially improving patient comfort and compliance. The protocol successfully addresses both skeletal and dental components of open bite malocclusion in growing patients.

DETAILED DESCRIPTION:
Detailed Description This prospective interventional study aimed to develop and evaluate a novel treatment protocol for skeletal open bite that eliminates the need for extraoral appliances while achieving comparable therapeutic outcomes. Skeletal open bite represents a challenging orthodontic condition characterized by increased vertical facial dimensions, divergent skeletal planes, and negative overbite.

Our treatment protocol combined two therapeutic approaches: (1) a modified open bite activator constructed with 3-4mm addition to the freeway space and relief in the anterior region, and (2) skeletal anchorage using mini-screws placed in the anterior region between lateral and canine teeth in both arches, connected by vertical intermaxillary elastics.

The open bite activator component functioned through multiple mechanisms: acting as a posterior bite block to inhibit posterior dentoalveolar eruption, serving as a tongue barrier to prevent tongue thrust between anterior teeth, and directing masticatory forces to the posterior segments. The anterior relief in the appliance allowed for uninhibited eruption of incisors. The vertical elastics between mini-screws provided controlled force (150g) to facilitate favorable rotational movements of the maxilla and mandible.

Cephalometric analyses included comprehensive skeletal angular measurements (SNA, SNB, ANB, Y Axis, SN/PP, GoGn/SN, PP/MP, gonial angle), skeletal linear measurements (N-Me, ANS-Me, Co-Go, S-Go), skeletal proportional measurements (Jarabak ratio), dentoalveolar angular measurements (U1-PP, interincisal angle, IMPA), and dentoalveolar linear measurements (overjet, overbite, U1-PP, U6-PP, L1-MP, L6-MP).

This treatment protocol demonstrates the potential to achieve effects similar to traditional approaches using posterior high-pull headgear and vertical chin cup, without compromising treatment outcomes. The significance of this approach lies in its ability to address a primary challenge in orthodontic treatment of growing patients with skeletal open bite: patient compliance and comfort, which often determines treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Growing individuals aged 12-14 years
* Diagnosis of skeletal open bite with GoGn/SN angle ≥36°
* Dentally reduced or negative overbite
* Ongoing growth and development (confirmed with hand-wrist radiographs)
* Good oral hygiene
* No prior orthodontic treatment or orthognathic surgery
* No systemic disease or craniofacial deformity
* Informed consent obtained from participant and parent/guardian

Exclusion Criteria:

* Presence of any craniofacial anomaly or systemic condition affecting craniofacial growth
* History of prior orthodontic treatment or jaw surgery
* Poor oral hygiene
* Non-compliance with appliance wear protocol
* Outside the age range of 12-14 years

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Change in GoGn/SN Angle (Mandibular Plane Angle) from Baseline to 12 Months | Baseline to 12 months post-treatment
  This outcome assesses the change in the mandibular plane angle (GoGn/SN) using lateral cephalometric radiographs taken at the beginning of treatment (T0) and after 12 months of therapy (T1). A decrease in the GoGn/SN angle indicates counterclockwise rotation of the mandible, which is a favorable skeletal change in the treatment of skeletal open bite. Measurements were performed using standardized digital cephalometric analysis software (Dolphin Imaging 11.95).

CONTACTS AND LOCATIONS:
Overall Officials: Elif Değirmenci, DDS, PhD, Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data (IPD), including cephalometric measurements, will be made available upon reasonable request to qualified researchers following publication. Requests should be directed to the corresponding author and will require a data use agreement.